CLINICAL TRIAL: NCT02679781
Title: Nasal Versus Oral Midazolam Sedation in Routine Pediatric Dental Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Avia Fux, pediatric dentist, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0678-15-HMO-CTIL
Record Dates: First submitted 2016-01-31; First posted 2016-02-10 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral sedation (Active Comparator): administration of 0.5mg/kg oral midazolam. During dental treatment 50% nitrous oxide/ 50% oxygen will be administered via nasal hood.
  Interventions: Drug: oral midazolam
- nasal sedation (Active Comparator): administration of 0.2mg/kg nasal midazolam. During dental treatment 50% nitrous oxide/ 50% oxygen will be administered via nasal hood.
  Interventions: Drug: nasal midazolam

INTERVENTIONS:
Drug: oral midazolam — administration of 0.5mg/kg oral midazolam. During dental treatment 50% nitrous oxide/ 50% oxygen will be administered via nasal hood.
  Other Names: oral dormicum
  Arms: oral sedation
Drug: nasal midazolam — administration of 0.2mg/kg nasal midazolam. During dental treatment 50% nitrous oxide/ 50% oxygen will be administered via nasal hood.
  Other Names: nasal dormicum
  Arms: nasal sedation

SUMMARY:
The general objective of the study is to compare the efficacy of administering midazolam orally as syrup versus nasally with nasal atomizer. The specific objectives are to measure: 1) acceptability of the medication, 2) effect on behavior, 3) time of onset, 4) maximum working time.

DETAILED DESCRIPTION:
* Prospective, parallel design
* Study and control group: 100 healthy children (ASA 1), ages: 2-6 years, uncooperative (Frankl 1-2), that needs at least two similar dental treatments. Exclusion criteria: enlarged tonsils (Brodsky's grading scale11 +3 = 50-75% airway obstruction, and +4 = >75% airway obstruction), upper respiratory tract infection or nasal discharge.
* Randomization: At the first appointment the subjects will assigned randomly to receive oral midazolam or nasal midazolam;
* Sedation: oral midazolam dose is 0.5mg/kg. Nasal midazolam dose is 0.2mg/kg. During treatment 50% nitrous oxide/ 50% oxygen will be administered via nasal hood.
* Acceptability of the medication: compliance in taking the medication will be assessed and recorded as: willingly, coaxed, forced, or failed (not administered).
* Behavior during dental treatment: Houpt scale measures behavior by rating sleep, movement, crying and overall behavior. The degree of alertness, movement and crying will be assessed before, during (every 5 min) and after the operative procedure. The rating will be done by one observer blind to the route of administration. This blind observer will also monitor the pulse and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* healthy children (ASA 1), uncooperative (Frankl 1-210), that needs at least two similar dental treatments.

Exclusion Criteria:

* enlarged tonsils (Brodsky's grading scale11 +3 = 50-75% airway obstruction, and +4 = >75% airway obstruction), upper respiratory tract infection or nasal discharge.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Fux-Noy A, Saadi Q, Shmueli A, Halperson E, Ram D, Moskovitz M. Parents' satisfaction and children's acceptance of nasal compared to oral midazolam for sedation in two consecutive pediatric dental treatments: a randomized controlled study. Front Dent Med. 2023 Dec 21;4:1296823. doi: 10.3389/fdmed.2023.1296823. eCollection 2023. PMID 39916898

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Sedation: administration of 0.5mg/kg oral midazolam.
- Nasal Sedation: administration of 0.2mg/kg nasal midazolam.
Period: Overall Study
Arm/Group | Oral Sedation | Nasal Sedation
Started | 37 | 33
Completed | 30 | 30
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — low cooperation, referral to treatment under general anesthesia | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Sedation | Nasal Sedation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Drop out- 10 were excluded from the analysis: seven due to lack of cooperation and referral to treatment under general anesthesia, six of whom received oral midazolam. Three participants did not attend the second treatment (one of them received oral midazolam).
  years | 4.25 (1.39) | 4.46 (1.25) | 4.36 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Drop out- 10 were excluded from the analysis: seven due to lack of cooperation and referral to treatment under general anesthesia, six of whom received oral midazolam. Three participants did not attend the second treatment (one of them received oral midazolam).
  Participants
    Female | 15 | 14 | 29
    Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Drop out- 10 were excluded from the analysis: seven due to lack of cooperation and referral to treatment under general anesthesia, six of whom received oral midazolam. Three participants did not attend the second treatment (one of them received oral midazolam).
  participants
    Israel | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Compliant With Oral or Nasal Midazolam Administration
Description: the compliance in taking the medication will be assessed at the time of administration by one of the investigators and recorded immediately as: willingly, coaxed, forced, or failed (not administered).
Time Frame: the compliance in taking the medication will be assessed at the time of administration and recorded immediately.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Sedation | Nasal Sedation
Number analyzed (Participants) | 30 | 30
Participants
  willingly | 11 | 4
  coaxed | 14 | 18
  forced | 5 | 8

2. Secondary Outcome: Behavior During Dental Treatment
Description: the effect of oral or nasal midazolam on behaviour will be assessed by blind observer using Houpt scale. Houpt scale measures behavior by rating overall behavior. the scale is 1 to 6, higher score mean a better behavior.
  1. = Aborted, no treatment rendered.
  2. = Poor, treatment interrupted, only partial treatment was completed 3= Fair, treatment interrupted but eventually completed 4= Good, difficult but all treatment was performed 5= Very good, some limited crying or movement 6= Excellent, no crying or movement
Time Frame: the effect of oral or nasal midazolam on behaviour will be assessed during dental treatment.The length of each treatment is estimated as 30-45 minutes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Sedation | Nasal Sedation
Number analyzed (Participants) | 30 | 30
score on a scale | 5.17 (0.79) | 4.80 (0.80)

ADVERSE EVENTS:
Time Frame: From administering the medication until recovery from sedation- at least 2 hours for each patient
Arm/Group | Oral Sedation | Nasal Sedation
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/33
Other Adverse Events (participants affected / at risk) | 0/37 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT02679781/Prot_SAP_000.pdf